CLINICAL TRIAL: NCT02934620
Title: Promoting CSD500 Use Among Women in Established Relationships
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Ministry of Health, Vietnam (Other Government); University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Maria F. Gallo, PhD, Associate Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2015H0242
Record Dates: First submitted 2016-10-10; First posted 2016-10-17 (Estimated); Results first posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-10

CONDITIONS: PSA; Unprotected Sex
Keywords: pregnancy; condom; HIV; sexually transmitted infections
MeSH Terms: conditions — Unsafe Sex; Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CSD500 Condom (Experimental): Receive CSD500 condoms with condom counseling to use them for sexual pleasure.
  Interventions: Device: CSD500 Condom; Behavioral: Condom Counseling
- Standard Condom (Active Comparator): Receive the standard condom with condom counseling to use them for pregnancy and disease prevention.
  Interventions: Device: Standard Condom; Behavioral: Condom Counseling

INTERVENTIONS:
Device: CSD500 Condom — CSD500 is a commercial condom that complies fully with the requirements of ISO 4074, the international standard for male latex condoms. The product is designed to increase sexual pleasure.
  Other Names: Blue Diamond
  Arms: CSD500 Condom
Device: Standard Condom — The standard condom is a standard condom in Vietnam at the time of the study. It is provided for pregnancy and disease prevention.
  Arms: Standard Condom
Behavioral: Condom Counseling — The intervention arm will receive counseling that briefly addresses condom's dual protection against pregnancy and HIV/STI but that otherwise emphasizes the potential for increased sexual pleasure with CSD500 use. Counseling to this arm also will include CSD500-specific instructions, such as the need to briefly massage the gel inside the condom teat onto the penis head after donning the condom and to not use multiple condoms within a 24-hour period. The control arm will receive standard counseling to use condoms for pregnancy and disease prevention without receiving any messages about the use of condoms for sexual pleasure.

SUMMARY:
Globally, women in established relationships remain at risk for unintended pregnancy and sexually transmitted infections (STIs), including HIV. In Vietnam, the location of the proposed research, unmet need for contraception is substantial as reflected in the nation's high abortion ratio. Married women account for about one-third of HIV cases in Vietnam, and among this group, most were exposed to the virus through sexual activity with their husband. Condoms will remain crucial for prevention for some time to come. Sustained condom use, however, is notoriously difficult to achieve. A key barrier to the consistent use of condoms is their effect on sexual pleasure. Although sexual pleasure is a primary motivation for engaging in sex and is an integral part of overall sexual health, most programs to improve sexual health operate within a pregnancy and disease-prevention paradigm. A new condom, CSD500, containing an erectogenic drug was developed for use among healthy couples to improve sexual pleasure by increasing penile firmness, size and erection duration. The overall objective of the proposed two-arm randomized trial is to test whether promoting the novel condom CSD500 for improved sexual pleasure results in couples having less unprotected vaginal sex. Investigators will measure the occurrence of unprotected vaginal sex by testing women's vaginal fluid for the presence of prostate-specific antigen (PSA), an objective, biological marker of recent semen exposure. Investigators will randomize 500 adult, heterosexual, monogamous couples, comprised of a total of 1000 individuals, in Thanh Hoa province, Vietnam to receive either CSD500 for sexual pleasure or the standard condom currently provided only for pregnancy and disease prevention to patients during routine care. Study staff will interview female participants at enrollment and after 2, 4, and 6 months and their male partners at the 6-month visit. Study clinicians will sample vaginal fluid from female participants at all visits to test for the presence of PSA.

DETAILED DESCRIPTION:
This randomized controlled trial will test whether promoting the novel condom CSD500 (Futura Medical Developments; Surrey, UK) for improved sexual pleasure results in couples having less unprotected vaginal sex - measured with a biological marker of recent semen exposure - compared to the promotion of a standard condom for disease and pregnancy prevention. CSD500 contains an erectogenic drug and was developed to improve sexual pleasure by increasing penile firmness, size, and erection duration.

Investigators will recruit eligible, monogamous, heterosexual couples at Thanh Hoa Provincial Centre of Reproductive Health in Vietnam to participate in a randomized controlled trial (RCT) of two balanced arms of approximately 250 heterosexual couples each, for a total of 500 couples, comprised of 1000 individuals. At enrollment and at three follow-up visits scheduled at 2, 4 and 6 months after enrollment, study staff will provide condom counseling, will collect vaginal swabs to test for the semen biomarker, prostate-specific antigen (PSA), and will administer a questionnaire to the female participants on their demographics, sexual and condom-related attitudes and practices, including sexual pleasure and perceptions of partner's sexual pleasure. Although the intervention is directed to the women, couples will be enrolled to ensure that the male partners consent to CSD500 use. After enrollment, male participants will not participate in study visit activities, including data collection, until the time of their female partner's final 6-month visit. Because of the differences in counseling messages, participants and study staff at the site cannot be blinded to arm assignment.

ELIGIBILITY:
Inclusion Criteria (for women):

* Not currently using a modern contraceptive method other than condoms or intending to start using a modern contraceptive method other than condoms in the next 6 months;
* Willing to use assigned study condoms as the sole method of contraception for the next six months;
* Not breastfeeding;
* Not known to be pregnant;
* Want to avoid pregnancy for at least the next six months; and
* Be in a monogamous relationship for at least the past six months with her current male partner.

Exclusion Criteria (for couples):

Couples are ineligible for study participation if either person in the couple is known to be HIV-positive or has any of the following contraindications to CSD500 use:

* History of low blood pressure or heart condition;
* Current use of medication for anemia, blood pressure, erectile dysfunction, migraines, headaches or glaucoma;
* Inflamed or broken skin that the condom could come into contact with; or
* Latex allergy or sensitivity.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1000 (Actual)
Dates: Start 2017-06-09 (Actual); Primary Completion 2020-02-19 (Actual); Study Completion 2020-02-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Gallo, PhD, Principal Investigator — Ohio State University; John Casterline, PhD, Principal Investigator — Ohio State University; Rebecca Andridge, PhD, Principal Investigator — Ohio State University; Marcia Hobbs, PhD, Principal Investigator — University of North Carolina; Nghia Nguyen, MD, PhD, Principal Investigator — Ministry of Health, Vietnam
Locations (1):
- Thanh Hoa Provincial Centre of Reproductive Health, Thanh Hóa, Thanh Hóa Province, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nguyen NC, Luong TN, Le VT, Hobbs M, Andridge R, Casterline J, Gallo MF. Effectiveness of erectogenic condom against semen exposure among women in Vietnam: Randomized controlled trial. PLoS One. 2022 Feb 17;17(2):e0263503. doi: 10.1371/journal.pone.0263503. eCollection 2022. PMID 35176037

RESULTS

PARTICIPANT FLOW:
Groups:
- CSD500 Condom - Female Participants; CSD500 Condom- Male Partners: Male and female partners were enrolled at together as a couple in the study.
  Receive CSD500 condoms with condom counseling to use them for sexual pleasure.
  CSD500 Condom: CSD500 is a commercial condom that complies fully with the requirements of ISO 4074, the international standard for male latex condoms. The product is designed to increase sexual pleasure.
  Condom Counseling: The intervention arm will receive counseling that briefly addresses condom's dual protection against pregnancy and HIV/STI but that otherwise emphasizes the potential for increased sexual pleasure with CSD500 use. Counseling to this arm also will include CSD500-specific instructions, such as the need to briefly massage the gel inside the condom teat onto the penis head after donning the condom and to not use multiple condoms within a 24-hour period. The control arm will receive standard counseling to use condoms for pregnancy and disease prevention without receiving any messages about the use of condoms for sexual pleasure.
- Standard Condom - Female Participants; Standard Condom - Male Partners: Male and female partners were enrolled at together as a couple in the study.
  Receive the standard condom with condom counseling to use them for pregnancy and disease prevention.
  Standard Condom: The standard condom is a standard condom in Vietnam at the time of the study. It is provided for pregnancy and disease prevention.
  Condom Counseling: The intervention arm will receive counseling that briefly addresses condom's dual protection against pregnancy and HIV/STI but that otherwise emphasizes the potential for increased sexual pleasure with CSD500 use. Counseling to this arm also will include CSD500-specific instructions, such as the need to briefly massage the gel inside the condom teat onto the penis head after donning the condom and to not use multiple condoms within a 24-hour period. The control arm will receive standard counseling to use condoms for pregnancy and disease prevention without receiving any messages about the use of condoms for sexual pleasure.
Period: Baseline Visit
Arm/Group | CSD500 Condom - Female Participants | Standard Condom - Female Participants | CSD500 Condom- Male Partners | Standard Condom - Male Partners
Started | 248 | 252 | 248 | 252
Completed | 248 | 252 | 248 | 252
Not Completed | 0 | 0 | 0 | 0
Period: 2-month Visit
Arm/Group | CSD500 Condom - Female Participants | Standard Condom - Female Participants | CSD500 Condom- Male Partners | Standard Condom - Male Partners
Started | 248 | 252 | 0 (Male partners were not asked to complete a 2-month visit.) | 0 (Male partners were not asked to complete a 2-month visit.)
Completed | 233 | 228 | 0 | 0
Not Completed | 15 | 24 | 0 | 0
Period: 4-month Visit
Arm/Group | CSD500 Condom - Female Participants | Standard Condom - Female Participants | CSD500 Condom- Male Partners | Standard Condom - Male Partners
Started | 248 (Our study procedures allowed female participants to attend the 4-month visit even if they had not attended the 2-month visit.) | 252 (Our study procedures allowed female participants to attend the 4-month visit even if they had not attended the 2-month visit.) | 0 (Male partners were not asked to complete a 4-month visit.) | 0 (Male partners were not asked to complete a 4-month visit.)
Completed | 228 | 220 | 0 | 0
Not Completed | 20 | 32 | 0 | 0
Period: 6-month Visit
Arm/Group | CSD500 Condom - Female Participants | Standard Condom - Female Participants | CSD500 Condom- Male Partners | Standard Condom - Male Partners
Started | 248 (Our study procedures allowed female participants to attend the 6-month visit even if they had not attended the 2-month and/or 4-month visit.) | 252 (Our study procedures allowed female participants to attend the 6-month visit even if they had not attended the 2-month and/or 4-month visit.) | 248 | 252
Completed | 234 | 239 | 230 | 238
Not Completed | 14 | 13 | 18 | 14

BASELINE CHARACTERISTICS:
Groups:
- CSD500 Condom - Male Participants: Male and female partners were enrolled at together as a couple in the study.
  Receive CSD500 condoms with condom counseling to use them for sexual pleasure.
  CSD500 Condom: CSD500 is a commercial condom that complies fully with the requirements of ISO 4074, the international standard for male latex condoms. The product is designed to increase sexual pleasure.
  Condom Counseling: The intervention arm will receive counseling that briefly addresses condom's dual protection against pregnancy and HIV/STI but that otherwise emphasizes the potential for increased sexual pleasure with CSD500 use. Counseling to this arm also will include CSD500-specific instructions, such as the need to briefly massage the gel inside the condom teat onto the penis head after donning the condom and to not use multiple condoms within a 24-hour period. The control arm will receive standard counseling to use condoms for pregnancy and disease prevention without receiving any messages about the use of condoms for sexual pleasure.
- Standard Condom - Male Participants: Male and female partners were enrolled at together as a couple in the study.
  Receive the standard condom with condom counseling to use them for pregnancy and disease prevention.
  Standard Condom: The standard condom is a standard condom in Vietnam at the time of the study. It is provided for pregnancy and disease prevention.
  Condom Counseling: The intervention arm will receive counseling that briefly addresses condom's dual protection against pregnancy and HIV/STI but that otherwise emphasizes the potential for increased sexual pleasure with CSD500 use. Counseling to this arm also will include CSD500-specific instructions, such as the need to briefly massage the gel inside the condom teat onto the penis head after donning the condom and to not use multiple condoms within a 24-hour period. The control arm will receive standard counseling to use condoms for pregnancy and disease prevention without receiving any messages about the use of condoms for sexual pleasure.
- Total: Total of all reporting groups
Arm/Group | CSD500 Condom - Female Participants | Standard Condom - Female Participants | CSD500 Condom - Male Participants | Standard Condom - Male Participants | Total
Number analyzed (Participants) | 248 | 252 | 248 | 252 | 1000
Age, Categorical [Count of Participants; unit: Participants] — Population: Age of male partners was not collected.
  Participants
    number analyzed (Participants) | 248 | 252 | 0 | 0 | 500
    <=18 years | 0 | 0 |  |  | 0
    Between 18 and 65 years | 248 | 252 |  |  | 500
    >=65 years | 0 | 0 |  |  | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Age of male partners was not collected.
  Years
    number analyzed (Participants) | 248 | 252 | 0 | 0 | 500
    (all) | 33.9 (5.3) | 34.3 (5.5) |  |  | 34.1 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 248 | 252 | 0 | 0 | 500
  Male | 0 | 0 | 248 | 252 | 500
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 248 | 252 | 248 | 252 | 1000
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Vietnam | 248 | 252 | 248 | 252 | 1000

OUTCOME MEASURES:

1. Primary Outcome: Number of Female Participants With Positive PSA at 2-Month Visit
Description: A double-headed vaginal swab is collected for each female participant to assess for PSA positivity.
Time Frame: Vaginal swab collected at 2-month follow-up visit
Population: Intent-to-treat
Measure: Count of Participants; unit: Participants
Groups:
- CSD500 Condom - Female Participants: Receive CSD500 condoms with condom counseling to use them for sexual pleasure.
  CSD500 Condom: CSD500 is a commercial condom that complies fully with the requirements of ISO 4074, the international standard for male latex condoms. The product is designed to increase sexual pleasure.
  Condom Counseling: The intervention arm will receive counseling that briefly addresses condom's dual protection against pregnancy and HIV/STI but that otherwise emphasizes the potential for increased sexual pleasure with CSD500 use. Counseling to this arm also will include CSD500-specific instructions, such as the need to briefly massage the gel inside the condom teat onto the penis head after donning the condom and to not use multiple condoms within a 24-hour period. The control arm will receive standard counseling to use condoms for pregnancy and disease prevention without receiving any messages about the use of condoms for sexual pleasure.
- Standard Condom - Female Participants: Receive the standard condom with condom counseling to use them for pregnancy and disease prevention.
  Standard Condom: The standard condom is a standard condom in Vietnam at the time of the study. It is provided for pregnancy and disease prevention.
  Condom Counseling: The intervention arm will receive counseling that briefly addresses condom's dual protection against pregnancy and HIV/STI but that otherwise emphasizes the potential for increased sexual pleasure with CSD500 use. Counseling to this arm also will include CSD500-specific instructions, such as the need to briefly massage the gel inside the condom teat onto the penis head after donning the condom and to not use multiple condoms within a 24-hour period. The control arm will receive standard counseling to use condoms for pregnancy and disease prevention without receiving any messages about the use of condoms for sexual pleasure.
Arm/Group | CSD500 Condom - Female Participants | Standard Condom - Female Participants
Number analyzed (Participants) | 233 | 228
Participants | 18 | 20

2. Primary Outcome: Number of Female Participants With Positive PSA at 4-Month Visit
Description: A double-headed vaginal swab is collected for each female participant to assess for PSA positivity.
Time Frame: Vaginal swab collected at 4-month follow-up visit
Measure: Count of Participants; unit: Participants
Arm/Group | CSD500 Condom - Female Participants | Standard Condom - Female Participants
Number analyzed (Participants) | 228 | 220
Participants | 12 | 12

3. Primary Outcome: Number of Female Participants With Positive PSA at 6-Month Visit
Description: A double-headed vaginal swab is collected for each female participant to assess for PSA positivity.
Time Frame: Vaginal swab collected at 6-month follow-up visit
Measure: Count of Participants; unit: Participants
Arm/Group | CSD500 Condom | Standard Condom
Number analyzed (Participants) | 234 | 239
Participants | 17 | 14

4. Secondary Outcome: Number of Female Participants With Self-reported Condomless Sex at 2-month Follow-up Visit
Description: Investigators will compare frequency of self-reports of recent sex without a condom between the two arms of female participants.
Time Frame: Measured at 2-month follow-up visit
Population: Intent-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | CSD500 Condom - Female Participants | Standard Condom - Female Participants
Number analyzed (Participants) | 233 | 227
Participants | 8 | 22

5. Secondary Outcome: Quality of Sexual Experience (QSE) Scale Scores Among Participants at 6-month Visit
Description: The Quality of Sexual Experience Scale was modified to add a question about pleasure related to the act's duration. The scale will be used to evaluate the effects of CSD500 provision on women and men's reports of sexual pleasure compared to the standard condom. The scale ranges from 0-7 points with a higher score indicating a higher-quality experience.
Time Frame: Measured among participants at at 6-month follow-up visit
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- CSD500 Condom - Male Participants: Receive CSD500 condoms with condom counseling to use them for sexual pleasure.
  CSD500 Condom: CSD500 is a commercial condom that complies fully with the requirements of ISO 4074, the international standard for male latex condoms. The product is designed to increase sexual pleasure.
  Condom Counseling: The intervention arm will receive counseling that briefly addresses condom's dual protection against pregnancy and HIV/STI but that otherwise emphasizes the potential for increased sexual pleasure with CSD500 use. Counseling to this arm also will include CSD500-specific instructions, such as the need to briefly massage the gel inside the condom teat onto the penis head after donning the condom and to not use multiple condoms within a 24-hour period. The control arm will receive standard counseling to use condoms for pregnancy and disease prevention without receiving any messages about the use of condoms for sexual pleasure.
- Standard Condom - Male Participants: Receive the standard condom with condom counseling to use them for pregnancy and disease prevention.
  Standard Condom: The standard condom is a standard condom in Vietnam at the time of the study. It is provided for pregnancy and disease prevention.
  Condom Counseling: The intervention arm will receive counseling that briefly addresses condom's dual protection against pregnancy and HIV/STI but that otherwise emphasizes the potential for increased sexual pleasure with CSD500 use. Counseling to this arm also will include CSD500-specific instructions, such as the need to briefly massage the gel inside the condom teat onto the penis head after donning the condom and to not use multiple condoms within a 24-hour period. The control arm will receive standard counseling to use condoms for pregnancy and disease prevention without receiving any messages about the use of condoms for sexual pleasure.
Arm/Group | CSD500 Condom - Female Participants | Standard Condom - Female Participants | CSD500 Condom - Male Participants | Standard Condom - Male Participants
Number analyzed (Participants) | 233 | 228 | 229 | 237
score on a scale | 5.27 (0.84) | 277 (5.13) | 5.48 (0.79) | 5.27 (0.66)

6. Secondary Outcome: Quality of Sexual Experience (QSE) Scale Scores Among Female Participants at 2-month Visit
Description: The Quality of Sexual Experience Scale was modified to add a question about pleasure related to the act's duration. The scale will be used to evaluate the effects of CSD500 provision on women's reports of sexual pleasure compared to the standard condom. The scale ranges from 0-7 points with a higher score indicating a higher-quality experience.
Time Frame: Measured among female participants at at 2-month follow-up visit
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Standard Condoms - Female Participants: Receive the standard condom with condom counseling to use them for pregnancy and disease prevention.
  Standard Condom: The standard condom is a standard condom in Vietnam at the time of the study. It is provided for pregnancy and disease prevention.
  Condom Counseling: The intervention arm will receive counseling that briefly addresses condom's dual protection against pregnancy and HIV/STI but that otherwise emphasizes the potential for increased sexual pleasure with CSD500 use. Counseling to this arm also will include CSD500-specific instructions, such as the need to briefly massage the gel inside the condom teat onto the penis head after donning the condom and to not use multiple condoms within a 24-hour period. The control arm will receive standard counseling to use condoms for pregnancy and disease prevention without receiving any messages about the use of condoms for sexual pleasure.
Arm/Group | CSD500 Condom - Female Participants | Standard Condoms - Female Participants
Number analyzed (Participants) | 233 | 227
score on a scale | 5.27 (0.84) | 5.13 (0.72)

7. Secondary Outcome: Quality of Sexual Experience (QSE) Scale Scores Among Female Participants at 4-month Visit
Description: as for outcome 6
Time Frame: Measured among female participants at at 4-month follow-up visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CSD500 Condom - Female Participants | Standard Condom - Female Participants
Number analyzed (Participants) | 226 | 220
score on a scale | 5.20 (0.71) | 5.07 (0.70)

8. Secondary Outcome: Number of Female Participants With Self-reported Condomless Sex at 4-month Follow-up Visit
Description: as for outcome 4
Time Frame: Measured at 4-month follow-up visit
Population: Intent-to-treat
Measure: Count of Participants; unit: Participants
Groups:
- Standard Condom- Female Participants: Receive the standard condom with condom counseling to use them for pregnancy and disease prevention.
  Standard Condom: The standard condom is a standard condom in Vietnam at the time of the study. It is provided for pregnancy and disease prevention.
  Condom Counseling: The intervention arm will receive counseling that briefly addresses condom's dual protection against pregnancy and HIV/STI but that otherwise emphasizes the potential for increased sexual pleasure with CSD500 use. Counseling to this arm also will include CSD500-specific instructions, such as the need to briefly massage the gel inside the condom teat onto the penis head after donning the condom and to not use multiple condoms within a 24-hour period. The control arm will receive standard counseling to use condoms for pregnancy and disease prevention without receiving any messages about the use of condoms for sexual pleasure.
Arm/Group | CSD500 Condom - Female Participants | Standard Condom- Female Participants
Number analyzed (Participants) | 227 | 220
Participants | 17 | 12

9. Secondary Outcome: Number of Female Participants With Self-reported Condomless Sex at 6-month Follow-up Visit
Description: as for outcome 4
Time Frame: Measured at 6-month follow-up visit
Population: Intent-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | CSD500 Condom - Female Participants | Standard Condom - Female Participants
Number analyzed (Participants) | 231 | 238
Participants | 16 | 14

ADVERSE EVENTS:
Time Frame: 6 months
Description: The number of participants at risk for all the adverse event terms are less than the **Total** number of participants at risk for other adverse events in both arms. This is due to missing data for some survey items. If the survey item did not have a response recorded, we did not include the participant in the number at risk.
  Other (Not Including Serious) Adverse Events were not monitored/assessed For "Male Partners" Arm/Groups.
Groups:
- Standard Condom -Male Participants: Receive the standard condom with condom counseling to use them for pregnancy and disease prevention.
  Standard Condom: The standard condom is a standard condom in Vietnam at the time of the study. It is provided for pregnancy and disease prevention.
  Condom Counseling: The intervention arm will receive counseling that briefly addresses condom's dual protection against pregnancy and HIV/STI but that otherwise emphasizes the potential for increased sexual pleasure with CSD500 use. Counseling to this arm also will include CSD500-specific instructions, such as the need to briefly massage the gel inside the condom teat onto the penis head after donning the condom and to not use multiple condoms within a 24-hour period. The control arm will receive standard counseling to use condoms for pregnancy and disease prevention without receiving any messages about the use of condoms for sexual pleasure.
Arm/Group | CSD500 Condom - Female Participants | Standard Condom - Female Participants | CSD500 Condom - Male Participants | Standard Condom -Male Participants
All-Cause Mortality (participants affected / at risk) | 0/248 | 0/252 | 0/248 | 0/252
Serious Adverse Events (participants affected / at risk) | 0/248 | 0/252 | 0/248 | 0/252
Other Adverse Events (participants affected / at risk) | 68/240 | 2/240 | 0/0 | 0/0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | CSD500 Condom - Female Participants (N=240) | Standard Condom - Female Participants (N=240) | CSD500 Condom - Male Participants (N=0) | Standard Condom -Male Participants (N=0)
Headaches at 2-month among Female Participants (General disorders) | 40/233 | 0/227 | 0 | 0
Headaches at 4-month among Female Participants (General disorders) | 32/227 | 0/220 | 0 | 0
Headaches at 6-month among Female Participants (General disorders) | 24/233 | 0/238 | 0 | 0
Dizziness at 2 months among Female Participants (General disorders) | 24/233 | 1/227 | 0 | 0
Dizziness at 4 months among Female Participants (General disorders) | 12/227 | 1/220 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-08-27): https://cdn.clinicaltrials.gov/large-docs/20/NCT02934620/Prot_SAP_000.pdf
  • Informed Consent Form (2017-01-31): https://cdn.clinicaltrials.gov/large-docs/20/NCT02934620/ICF_001.pdf